CLINICAL TRIAL: NCT00678015
Title: A Phase II Pharmacokinetic and Efficacy Study of Nordihydroguaiaretic Acid (NDGA) in Non-Metastatic Recurrent Prostate Cancer
Brief Title: Pharmacokinetic and Efficacy Study of Nordihydroguaiaretic Acid (NDGA) in Non Metastatic Recurrent Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per protocol - interim analysis showed no significant PSA declines among the first 12 patients after 3 cycles of treatment
Sponsor: University of California, San Francisco (Other)
Collaborators: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 075511
Record Dates: First submitted 2008-05-12; First posted 2008-05-15 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: NDGA; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Masoprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Nordihydroguaiaretic Acid (NDGA)

INTERVENTIONS:
Drug: Nordihydroguaiaretic Acid (NDGA) — NDGA 2000mg daily

SUMMARY:
This is a Phase II, single center study measuring the pharmacokinetic parameters of NDGA administration and assessing the proportion of patients who experience a 50% decline in PSA.

DETAILED DESCRIPTION:
This study is a phase II trial of NDGA in patients with hormone-sensitive non-metastatic prostate cancer with a pharmacokinetics component. The first six patients enrolled will be treated with a single 750 mg dose of oral NDGA on day -7 with measurement of pharmacokinetic parameters over eight hours after the dose, then begin treatment with 2000 mg of oral NDGA daily. Every four weeks, measurement of pharmacokinetic parameters at steady state will be done for all patients. All patients will continue dosing with NDGA and will be followed for PSA response and for safety. Measurement of pharmacokinetics for a 750 mg dose has been chosen to evaluate levels with the dosage that patients will be taking at one time point during the day (this is roughly one-third of the daily dose, which is administered in three divided doses).

ELIGIBILITY:
Inclusion Criteria:

* Rising prostate-specific antigen (PSA) value after local therapy with a PSA doubling time (PSADT) between 6 and 24 months (four or more readings at least two weeks apart within the last six months)
* Prior definitive therapy for prostate cancer consisting of one of the following:

  1. External beam radiotherapy with or without hormone therapy
  2. Brachytherapy with or without pelvic external beam radiation or hormone therapy
  3. Radical prostatectomy with or without adjuvant or salvage radiation therapy
* PSA > 1 ng/ml, which has risen serially on two determinations at least one week apart
* Progressive disease by "Phoenix" consensus definition for patients who have undergone primary radiation therapy (PSA nadir + 2 ng/mL)
* No metastatic disease
* Prior adjuvant or neoadjuvant androgen deprivation is permitted, provided:

  1. > 6 months since last day of effective androgen deprivation
  2. Testosterone > 250 ng/dL
  3. Patient is not on intermittent androgen deprivation
* Karnofsky performance status (KPS) of > 70%
* Liver Function Tests are within normal range
* Glycated hemoglobin (HgA1c) < 6%
* Patients must be four weeks from major surgery or radiotherapy to be eligible

Exclusion Criteria:

* Presence of another active malignancy other than prostate cancer, or treated squamous/basal cell carcinoma of the skin. Concomitant medical condition which would make it undesirable, in the physician's opinion, for the patient to participate in the protocol or would jeopardize compliance with the protocol requirements
* Diabetes mellitus, unless diet-controlled
* Must be off saw palmetto, pomegranate juice, finasteride, or any herbal agent intended to lower PSA for > 4 weeks. Baseline PSADT calculation must occur off of these agents
* Patients may not have evidence of local-only recurrence of prostate cancer
* No history of liver disease, including Hepatitis B or C, alcoholic liver disease, or autoimmune liver disease. A prior history of Hepatitis A is allowed provided that baseline liver function tests are within normal limits
* Patients with castration resistant prostate cancer are ineligible (prostate cancer which has progressed on androgen deprivation therapy with a Luteinizing hormone-releasing hormone (LHRH)-agonist or orchiectomy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Friedlander TW, Weinberg VK, Huang Y, Mi JT, Formaker CG, Small EJ, Harzstark AL, Lin AM, Fong L, Ryan CJ. A phase II study of insulin-like growth factor receptor inhibition with nordihydroguaiaretic acid in men with non-metastatic hormone-sensitive prostate cancer. Oncol Rep. 2012 Jan;27(1):3-9. doi: 10.3892/or.2011.1487. Epub 2011 Oct 4. PMID 21971890

RESULTS

PARTICIPANT FLOW:
Groups:
- NDGA: Nordihydroguaiaretic Acid (NDGA) 2000mg given orally daily in 3 divided doses (750mg in the morning and in the evening, and 500mg at midday) over a 28-day cycle.
Period: Overall Study
Arm/Group | NDGA
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NDGA
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 67.5 [55 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response According to Consensus Criteria
Description: Participants who experienced a PSA decline of at least 50%, confirmed by a second PSA value 4 or more weeks later. The reference PSA for decline was a PSA measured within 2 weeks of beginning study treatment. If at most 1 PSA response was observed among the first 12 patients, then accrual would stop and the trial would close for futility.
Time Frame: Monthly, up to 29 months
Measure: Number; unit: participants
Arm/Group | NDGA
Number analyzed (Participants) | 12
participants | 0

2. Post Hoc Outcome: PSA Decline
Description: Number of participants experiencing PSA decline during the first 3 treatment cycles
Time Frame: Baseline; Monthly, up to 29 months after beginning treatment
Measure: Number; unit: participants
Arm/Group | NDGA
Number analyzed (Participants) | 12
participants | 7

3. Post Hoc Outcome: Change in Prostate Specific Antigen Doubling Time (PSADT)
Description: PSADT was calculated using the formula natural log 2 divided by the slope of the natural log of the PSA versus time. Pretreatment PSADT was calculated using a minimum of 3 values; end of study PSADT incorporated all measured PSA values on study starting Cycle 2-Day 1 until the patient was removed from the study.
Time Frame: Cycle 2 through end of treatment (up to 29 months)
Population: At the time of PSADT calculations, one participant was still on study at 29 months, and 11 participants' time on study had ranged from 2-19 months
Measure: Median (Full Range); unit: percentage change
Arm/Group | NDGA
Number analyzed (Participants) | 12
percentage change | 17 [-66 to 72]

4. Post Hoc Outcome: Disease Progression at End of Study
Description: End-of-study imaging was assessed for disease progression per Response Evaluation Criteria In Solid Tumors (RECIST) criteria: * Progressive Disease (PD)=At least a 20% increase in the sum of the largest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline, End of treatment (2-19 cycles)
Population: At the time of calculation, 1 patient was still on study after 29 cycles
Measure: Number; unit: participants
Arm/Group | NDGA
Number analyzed (Participants) | 11
participants | 0

ADVERSE EVENTS:
Time Frame: Monthly during study treatment, 2-33 months
Description: Patients were evaluated monthly for toxicity, which was graded according to common toxicity criteria (CTC) 3.0
Arm/Group | NDGA
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NDGA (N=12)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Cognitive disturbance (Psychiatric disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (12)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated Alkaline phosphatase (General disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 4 (4)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (General disorders) | 1 (1)
Nausea (General disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Elevated ALT (Hepatobiliary disorders) | 8 (8)
Elevated AST (Hepatobiliary disorders) | 6 (6)
Elevated bilirubin (Hepatobiliary disorders) | 3 (3)
Elevated CPK (Hepatobiliary disorders) | 1 (1)
Elevated GGT (Hepatobiliary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Per protocol - accrual was stopped early after a pre-planned interim analysis showed no significant PSA declines after 3 cycles of treatment among the first 12 patients enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes